CLINICAL TRIAL: NCT04778137
Title: The Study of Omalizumab (CMAB007 and Xolair) in Healthy Subjects to Compare the PK, PD and Safety
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taizhou Mabtech Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CMAB007-001
Record Dates: First submitted 2021-02-26; First posted 2021-03-02 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CMAB007 (Experimental): 75mg×2
  Interventions: Drug: Omalizumab
- Xolair (Active Comparator): 150mg
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: Omalizumab — Biological: CMAB007 Biological: Xolair

SUMMARY:
A phase 1, randomized, double-blind, parallel group, single-dose study to compare the pharmacokinetics, pharmacodynamics and safety of two formulations of Omalizumab (CMAB007 and Xolair) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject between the ages of 18 and 45 years.
* Subject with a body weight of ≥50 kg and ≤ 75kg and a BMI between 19.0~26.0 kg/m2 (both inclusive).

Exclusion Criteria:

* subject has a medical history and/or current presence of disease
* subject has undergone surgery within three months before signing the informed consent;
* Alcoholics or regular drinkers within 3 months before the test, i.e. those who drink more than 14 unites of alcohol per week (14 bottles of 360 ml beer or 630 ml spirits with 40% alcohol), or whose alcohol breath test is positive;
* Those who have used soft drugs within 3 months prior to signing the informed consent or hard drugs within 1 year prior the trial; those who have positive drug abuse test results;
* Those who smoke more than 10 cigarettes per day on average in the 6 months before signing the informed consent; or those who have positive nocotine results;
* Those who have a history of drug or food allergy, or who have special allergy history (asthma, urticaria, etc.); those who have allergic rhinitis, or are known to be allergic to any component of the test drug or latex (contained in the syringe needle cover);
* Those who drinking too much tea, coffee and/or caffeinated beverages (more than 8 cups, 1 cup =250 ml) every day;
* Those who have received any drug treatment (including prescription drugs, over-the-counter drugs, biological products, Traditional Chinese medicine, etc.) and health care products within 4 weeks befor signing the informed consent;
* Those who have a blood donation over 400 ml within 3 months, or 200 ml within 1 month before signing the informed consent, or plan to donate blood during the trail;
* Those who accept any biological drugs within 3 months, or anti-IgE biological drugs within 12 months before signing the informed consent;
* Those who plan to donate sperm within 6 months after the administration of the test drug;
* Participants in other clinical trails within 3 months before signing the informed consent;
* Any one of HIV antibody, HBsAg, HBeAg, HBcAg, HCV antibody and Treponerma pallidum antibody is positive;
* The results of medical examination (ECG, X-ray, B-ultrasonic, physical and laboratory examination) are clinical significant abnormalities according to the judgment of the researcher;
* Anti-nuclear antibody or fecal parasite test is positive;
* Those who have undergone surgery within 1 months before signing the informed consent, or plan to undergo surgery during the trail period;

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Outcome Measures [AUC0-inf] | up to day 106
  Area Under the Concentration-time Curve from Time zero to infinity (AUC0-inf) of CMAB007 and Xolair in healthy subjects.
Pharmacokinetic Outcome Measures [Cmax] | up to day 106
  Maximum serum concentration (Cmax) of CMAB007 and Xolair in healthy subjects.

SECONDARY OUTCOMES:
Pharmacokinetic Outcome Measures [Tmax] | up to day 106
  Time to Cmax (Tmax) of CMAB007 and Xolair in healthy subjects
Pharmacokinetic Outcome Measures [t1/2] | up to day 106
  Terminal half-life (t1/2) of CMAB007 and Xolair in healthy subjects
Pharmacokinetic Outcome Measures [λz] | up to day 106
  Terminal elimination rate constant (λz) of CMAB007 and Xolair in healthy subjects
Pharmacokinetic Outcome Measures [Apparent total body clearance (CL/F)] | up to day 106
  Apparent total body clearance (CL/F) of CMAB007 and Xolair in healthy subjects
Pharmacodynamics [IgE levels] | up to day 106
  Free IgE and total IgE levels (the sum of free and omalizumab-bound IgE) in the serum samples from subjects
Incidence of Treatment-Emergent Adverse Events [Safety] | up to day 106
  Treatment-Emergent Adverse Events (TEAEs) of CMAB007 and Xolair in healthy subjects
Pharmacokinetic Outcome Measures [AUC0-t] | up to day 106
  Area Under the concentration-time Curve from time zero to the last quantifiable concentration (AUC0-t) of CMAB007 and Xolair in healthy subjects.
Pharmacokinetic Outcome Measures [Vd/F] | up to day 106
  Apparent total distribution (Cd/F) of CMAB007 and Xolair in healthy subjects
Immunogenicity | up to day 106
  the Immunogenicity of CMAB007 and Xolair in healthy subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No